CLINICAL TRIAL: NCT06006182
Title: The Effects of Freeze-Dried Whole Grape Powder on Chronic Disease and Cardiovascular Risk Factors, Hunger, Satiety, and Body Composition in Free-Living People-a Pilot Study
Brief Title: The Effects of Freeze-Dried Whole Grape Powder on Chronic Disease and Cardiovascular Risk Factors-a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State Polytechnic University, Pomona (Other)
Collaborators: The California Table grape Commission (Other)
Responsible Party: Principal Investigator, Dr. Bonny Burns-Whitmore, RD, Professor/Researcher, California State Polytechnic University, Pomona
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 100060; 24-04-101 (Other: Agriculture Research Institute)
Record Dates: First submitted 2023-08-01; First posted 2023-08-23 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Healthy People
MeSH Terms: interventions — whole grape extract

STUDY DESIGN:
Intervention Model Description: The crossover design can differentiate the diet treatment effect from other effects like secular trends and differential carryover, utilizes a perfect control (the experimental subject is the same person as the control), the subjects will experience all treatments (best for subject retention), and this study design does not require very many participants to provide adequate study power. The alpha is set at 0.05, and the power at 80%. Based on the calculations, the required number of participants in order to see a difference is 22. However, since a crossover study assumes a >20% dropout rate, the minimum of 20% is added to the minimum sample size of 22 at an alpha of 0.05 and a power of 80 (14). Therefore, we will be recruiting 30 adults. Since a parallel design would require 58 per treatment group (total=116), it was determined by the PIs that the crossover design was the best design for this study.
Who Masked: Participant
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A-Grape Powder then Placebo (Experimental): Group A block will be the Grape Powder for the first 8 weeks, and then after the washout period, they will begin the Placebo. The experimental Grape Powder is a food-it is simply freeze-dried grape powder
  Interventions: Other: Grape Powder
- Group B-Placebo-then Grape Powder (Placebo Comparator): Group B block will be the Placebo for the first 8 weeks, and then after the washout period, they will begin the Grape Powder
  Interventions: Other: Grape Powder

INTERVENTIONS:
Other: Grape Powder — Freeze-dried grape powder

SUMMARY:
Cardiovascular disease (CVD) is responsible for 1 out of every 5 deaths, is the number one killer of Americans, killing about 700K US adults per year (1). Our proposed research is a clinical trial that will determine the effects of feeding California freeze-dried grapes (which are directly comparable to fresh table grapes), on cardiovascular and chronic disease risk factors, namely, blood glucose and lipids (total cholesterol, LDL, HDL, and triacylglycerides), electrolyte and blood indicators (such as sodium, calcium, potassium, etc.), c-reactive protein (hs-CRP) and tumor necrosis factor alpha (TNF-alpha) (measures of inflammation and CVD risk), body composition (body weight, body fat percentage, lean tissue weight, body water amount and Kcal requirement to maintain body composition status), and blood pressure (BP) in 30 adults. The investigators will test satiety and hunger to see if grape antioxidants decrease both, implying that there will be a decrease in caloric intake and result in body composition improvements.

DETAILED DESCRIPTION:
METHODOLOGY/EXPERIMENTAL DESIGN-CROSSOVER

We plan to test the effects of feeding grapes (using the supplied freeze-dried grape powder from the California Table Grape Commission) in subjects aged 18 years of age or older. This study will be done in a free-living population, using a double-blinded randomized clinical trial (RCT) crossover study design at California Polytechnic University, Pomona

There will be a 3-month recruitment and screening period in which approximately 60 persons will be screened. There will be two 8-week randomized diet periods (to either Group A or B) separated by a washout period. Subjects will follow each of the randomly assigned diets: Freeze-Dried Grapes (Experimental/Treatment) for 8 weeks or Freeze-Dried Control (supplied by California Table Grape Commission), once a day for 8 weeks. The control diet-consumed during one of the treatment arm periods-will consist of the person's normal (habitual) diet with the absence of grapes in any form (including alcohol) and a grape-look alike placebo. The experimental diet will consist of the normal (habitual) diet of each subject, with the addition of the freeze-dried grapes in a 6 oz glass of water per day and the absence of grapes in any form. There will be a 5-8 week washout period between the two treatments.

Blood drawings, BP, hs-CRP and TNF-alpha, and body composition measurements will be performed on each subject at week 0, and after 8 weeks of each period arms. A phlebotomist at the California Polytechnic University, Pomona (CPP) Student Health Center, will draw the blood samples. An independent laboratory will analyze the coded blood samples for triglycerides, glucose, hs-CRP and TNF-alpha, total blood cholesterol, LDL, and HDL cholesterol levels.

Body composition will be measured using a Tanita Bioimpedance scale (T-310) and blood pressure will be taken with the OMRON blood pressure monitor.

As well, three 24-hour randomized diet recalls will be administered during each treatment to obtain information regarding the subject's diet and adherence to the diet protocol, and ESHA Research Food Processor will be used to analyze the diet. Adherence to the assigned diets will be assessed using an Unusual Diet Diary, which is filled out by the participant when unusual quantities of foods or accidental grape consumption occurs, medical treatment is required, pharmaceuticals/antioxidant supplements are consumed, or the participant exercises to excess. Visual Analog Questionnaires will be used to determine satiety and hunger during both study periods the day after the diet recall is obtained.

Subjects will pick up their study material allotment every week from the PI's office which is in room #119 in the Don B. Huntley College of Agriculture at Cal Poly Pomona. After Informed Consent is obtained, subjects will be instructed on how to mix the freeze-dried powder into the water as per the California Table Grape protocol.

Timetable The study timeline is 1 year, (includes subject recruitment, the study duration, laboratory analyses, and 2-3 months to organize and analyze the data, provide a report to the funders, and publish the results). The study, after obtaining participants, will commence at the beginning of August 2023, and end July 31, 2024. The two Co-PIs, two graduate students and 4 undergraduate students will conduct this study. The undergraduate students will help in recruitment and retention as well as performing, input and analysis of the 24-hour recalls in the ESHA software, Tanita measurements, passing out the subject's allocations, and tabulating the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy adults
* Attend school at or are employed by Cal Poly Pomona
* Not sensitive or allergic to grapes or grape products.
* Must be available 8 weeks during both Fall (2023) and Spring (2024) semesters.

Exclusion Criteria:

* Do not attend or are not employed by Cal Poly Pomona
* Smokers
* Pregnancy
* Any allergies to or dislike of grapes
* Cross-reactive allergies to grapes such as any of the following: peach, tree nuts, mustard, mulberry, cabbage, figs, kiwi, bananas, melon, apple, cherries, strawberries
* Thyroid disease
* Insulin dependent diabetes
* Non-insulin dependent diabetes
* Cancer
* Cardiovascular diseases
* Body piercings that cannot be removed
* Implanted devices
* Not available for 8 weeks during both (2023) and Spring (2024) semesters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Risk Blood Indicators | 8 weeks for placebo, 8 weeks for grape arms
  To determine if grape consumption changes (mg/d) fasting blood glucose, total cholesterol, low density lipoproteins, high density lipoproteins, and triacylglycerides

SECONDARY OUTCOMES:
Body Composition Changes-Percent Body Fat | 8 weeks for placebo, 8 weeks for grape arms
  To determine if grape consumption changes percent body fat.
Body Composition Changes-Body Water | 8 weeks for placebo, 8 weeks for grape arms
  To determine if grape consumption changes (Kg) body water.
Body Composition Changes-Lean Body Tissue | 8 weeks for placebo, 8 weeks for grape arms
  To determine if grape consumption changes (Kg) body lean tissue.
Inflammatory Factors-C-Reactive Protein | 8 weeks for placebo, 8 weeks for grape arms
  To determine if grape consumption changes inflammation as measured by changes (pg/mL) in C-reactive protein.
Inflammatory Factors-Tumor Necrosis Factor Alpha | 8 weeks for placebo, 8 weeks for grape arms
  To determine if grape consumption changes inflammation as measured by changes (mg/L) in tumor necrosis factor alpha
Blood Pressure | 8 weeks for placebo, 8 weeks for grape arms
  To determine if grape consumption changes (mm Hg) blood pressure.
Dietary Analysis-Obtain Diet Recalls | 8 weeks for placebo, 8 weeks for grape arms
  To obtain (3) 24-hour diet recalls per person in each treatment arm.
Dietary Analysis- Diet Intake | 3 times during the 8 weeks of each arm
  To assess changes in (g) dietary intake from the (3) 24-hour recalls in each treatment arm.
Dietary Analysis-Diet Antioxidants | 8 weeks for placebo, 8 weeks for grape arms
  To assess changes in (mg) dietary antioxidants consumed and antioxidant supplement use from the (3) 24-hour recalls.
Dietary Analysis-Diet Comparison | 8 weeks for placebo, 8 weeks for grape arms
  To assess changes in diet quality by comparing the placebo diet analyses with the grape diet analyses from the (3) 24-hour recalls.
High Blood Pressure Blood Indicators | 8 weeks for placebo, 8 weeks for grape arms
  To determine if grape consumption changes (mg/d) blood calcium, potassium and sodium.
Satiety | 3 times during the 8 weeks of each arm
  Using a visual analog scale, determine if grape consumption changes satiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Cal Poly Pomona, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share the data with other researchers.

REFERENCES:
- [Background] 1. Centers for Disease Control and Prevention, National Center for Health Statistics. About Multiple Cause of Death, 1999-2020. CDC WONDER Online Database website. Atlanta, GA: Centers for Disease Control and Prevention; 2022. Accessed January 14, 2023
- [Background] 2. Diabetes in Control. New and Information for Medical Professionals. Hyperglycemia Starts at 90mg.dL, That's Right Hyperglycemia. Online website. Accessed January 14, 2023
- [Background] Nelson RH. Hyperlipidemia as a risk factor for cardiovascular disease. Prim Care. 2013 Mar;40(1):195-211. doi: 10.1016/j.pop.2012.11.003. Epub 2012 Dec 4. PMID 23402469
- [Background] 4. Centers for Disease Control and Prevention. CDC 24/7: Saving Lives, Protecting People. Salt. Sodium, Potassium and Health. Online website. Accessed January 14, 2023.
- [Background] Arulselvan P, Fard MT, Tan WS, Gothai S, Fakurazi S, Norhaizan ME, Kumar SS. Role of Antioxidants and Natural Products in Inflammation. Oxid Med Cell Longev. 2016;2016:5276130. doi: 10.1155/2016/5276130. Epub 2016 Oct 10. PMID 27803762
- [Background] 6. National Center for Complementary and Integrative Health (NCCIH). Antioxidants: In Depth. https://nccih.nih.gov/health/antioxidants/introduction.htm. Online website. Accessed January 14, 2023.
- [Background] 7. USDA Oxygen Radical Absorbance Capacity (ORAC) of Selected Foods, Release 2 (2010). http://www.orac-info-portal.de/download/ORAC_R2.pdf Accessed January 12, 2024.
- [Background] Aune D, Giovannucci E, Boffetta P, Fadnes LT, Keum N, Norat T, Greenwood DC, Riboli E, Vatten LJ, Tonstad S. Fruit and vegetable intake and the risk of cardiovascular disease, total cancer and all-cause mortality-a systematic review and dose-response meta-analysis of prospective studies. Int J Epidemiol. 2017 Jun 1;46(3):1029-1056. doi: 10.1093/ije/dyw319. PMID 28338764
- [Background] Miller V, Mente A, Dehghan M, Rangarajan S, Zhang X, Swaminathan S, Dagenais G, Gupta R, Mohan V, Lear S, Bangdiwala SI, Schutte AE, Wentzel-Viljoen E, Avezum A, Altuntas Y, Yusoff K, Ismail N, Peer N, Chifamba J, Diaz R, Rahman O, Mohammadifard N, Lana F, Zatonska K, Wielgosz A, Yusufali A, Iqbal R, Lopez-Jaramillo P, Khatib R, Rosengren A, Kutty VR, Li W, Liu J, Liu X, Yin L, Teo K, Anand S, Yusuf S; Prospective Urban Rural Epidemiology (PURE) study investigators. Fruit, vegetable, and legume intake, and cardiovascular disease and deaths in 18 countries (PURE): a prospective cohort study. Lancet. 2017 Nov 4;390(10107):2037-2049. doi: 10.1016/S0140-6736(17)32253-5. Epub 2017 Aug 29. PMID 28864331
- [Background] 10. Mayo Clinic. Healthy Lifestyle. Nutrition and healthy eating. DASH diet: Healthy eating to lower your blood pressure. Online website. Accessed December 12, 2022.

DOCUMENTS (1):
  • Informed Consent Form (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT06006182/ICF_000.pdf